CLINICAL TRIAL: NCT00177164
Title: A Random Assignment,Parallel Group, Open Label Comparison of Clinical Outcomes and Resource Utilization Among Bipolar Disorder Patients Receiving Either Long Acting Injectable Risperidone Microspheres (Risperdal Consta® ) or Other Second Generation Oral Antipsychotic Agents: A 15 Month Study
Brief Title: Risperdal Consta for Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIS-PSY-405; Univ. Pittsburgh IRB #0403091
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Risperidone Consta - Long Acting Injection; Oral second generation antipsychotic agents
MeSH Terms: interventions — Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral Risperidone followed by Long acting Risperidone injections (Consta)
  Interventions: Drug: Injectable Risperidone (Consta) or oral antipsychotic
- 2 (Active Comparator): Oral second generation antipsychotic agents other than clozapine or risperidone (olanzapine, quetiapine, ziprasidone, aripiprazole)
  Interventions: Drug: Injectable Risperidone (Consta) or oral antipsychotic

INTERVENTIONS:
Drug: Injectable Risperidone (Consta) or oral antipsychotic — Injectable Risperidone (Consta) from 12.5 to 50 mg q 2 weeks
  Oral antipsychotic agents, olanzapine, quetiapine, ziprasidone, aripiprazole in doses approved in the US for bipolar disorder
  Other Names: Long actiing risperidone injection (Consta), oral risperidone (risperdal).; Olanzapine (Zyprexa), Quetiapine (Seroquel), Ziprasidone (Geodon), Aripiprazole (Ablify)

SUMMARY:
We recruited 50 consenting adult subjects with DSM-IV TR diagnoses of bipolar disorder who were about to initiate or switch their current antipsychotic agent. Only 48 patients (23 in the risperidone LAI group and 25 in the oral AAP group) contributed data to the assessments. Patients were titrated and cross-tapered during a 3 month titration and stabilization phase. They were followed for an additional 12 months. Clinical outcomes such as study drop out, adverse events, worsening of symptoms, crisis interventions, need for additional medication, hospitalizations etc. were evaluated from months 3 to 15. The numbers of clinical events (pooled) will be used to evaluate if the long acting injectable form of risperidone has an advantage over the oral second generation antipsychotic agents in terms of treatment continuity and clinical stability.

DETAILED DESCRIPTION:
OBJECTIVE:

To evaluate if a long acting injectable form of risperidone offers clinical advantages over comparison oral second generation antipsychotic agents following titration and stabilization in bipolar subjects. In keeping with current practice, it is expected the vast majority of patients will also be receiving either lithium or valproate or other anticonvulsants. Following the stabilization phase several clinical events will be evaluated for up to 15 months in the two treatment groups to examine differences in clinical outcomes between those receiving the injectable versus oral medicines.

RESEARCH PLAN:

We intend to recruit 50 consenting adult subjects with DSM-IV TR diagnoses of bipolar disorder who are about to initiate or to switch their antipsychotic agent. Patients will be titrated and cross-tapered during a 3 month titration and stabilization phase. Those who transition successfully and show some improvement will be followed for an additional 12 months. Clinical outcomes such as study drop out, adverse events, worsening of symptoms, crisis interventions, need for additional medication, hospitalizations etc. will be evaluated from months 3 to 15. The numbers of clinical events (pooled) will be used to evaluate if the long acting injectable form of risperidone has an advantage over the oral second generation antipsychotic agents in terms of treatment continuity and clinical stability.

METHODS:

An open design, but treatment to either the long acting risperidone or to the oral second generation antipsychotic agents is randomly assigned. A board independent of the day-to-day clinical events will code the primary clinical outcomes of interest without knowledge of treatment assignment. The board will be provided clinical summaries of these events without revealing the treatment assignment.

SIGNIFICANCE:

The use of a long acting injectable second generation antipsychotic agent may offer advantages of treatment continuity and adherence in bipolar patients permitting improved clinical stability and improved psychosocial and functional outcomes. Such stability is difficult to achieve in the face of frequent treatment discontinuations seen with oral agents. The improved tolerability of the second generation antipsychotic agents may change the perception of long acting injections. For instance, these agents are likely to be more acceptable to patients, families and clinicians and therefore likely be used much sooner in the treatment algorithms of bipolar patients than in the past. This study will provide a treatment effect size to statistically power future comparisons of long-acting injectable vs. oral antipsychotic agents in persons with bipolar disorder

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV - TR diagnoses of bipolar disorder (I or II or NOS).
* Age 18 to 70 years
* Men or women
* Any Ethnicity
* Currently receiving or willing to receive treatment at sites associated with the Western Psychiatric Institute and Clinic -University of Pittsburgh Medical Center (inpatient or ambulatory) or Mon Yough Community Services, Inc. or at Mayview State Hospital, Bridgeville, PA (inpatient)
* Able to provide competent and sign an informed consent document
* It is clinically appropriate in the eligible individual to consider antipsychotic treatment for at least 15 months (clinician and investigator determined)
* It is clinically appropriate to switch antipsychotic treatment to one of the second generation antipsychotic agents being evaluated in this study.
* There is no known contraindication for the use of either risperidone or for more than two of the antipsychotic agents being considered in the study (Investigator determined)
* At entry (at the screening visit, and just prior to randomization) Y-MRS (Young-Mania rating scale, Young et al., 1978) total score > 15 in bipolar disorder patients entering in a manic or mixed or hypomanic or NOS episode.
* Either life-time or current comorbid substance abuse or dependence is permitted (unless the Investigator and referring physician opines the substance abuse is likely to significantly interfere with either the diagnosis of the Axis I condition or to compromise patients safety due to withdrawal issues (Investigator determined).
* Screening physical and laboratory/EKG procedures are within acceptable limits

Exclusion Criteria:

* Actively suicidal or dangerous to others (Investigator opines that it is inappropriate to involve the potential subject in the study)
* Pregnant or lactating women
* Women in the reproductive age group who are not using any acceptable contraception (abstinence is not acceptable) or intend to become pregnant during the trial
* Subjects who are likely to face incarceration during the study duration (and for those already in the study, the continued participation of such subjects will be evaluated on a case-by-case basis)
* Patients currently receiving clozapine (or within six weeks prior to randomization) are ineligible for the study
* Subjects currently receiving a depot neuroleptic injectable agent, or within 2 injection cycles of receiving the injection prior to randomization.
* Allergy or serious side effects (for instance - neuroleptic malignant syndrome) to either risperidone or to more than two of the other second-generation antipsychotic agents that have been approved for use in the U.S.A. (olanzapine, quetiapine, ziprasidone, aripiprazole-per investigator and referring clinician).
* Treatment resistance to either risperidone, or to more than two of the other antipsychotic agents in this trial (olanzapine, quetiapine, ziprasidone, aripiprazole).
* This is the first episode of mania, mixed or hypomania for patients.
* Current (or within one month prior to randomization) participation in an investigational drug/device study.
* Currently participating in another study that would confound the present study objectives (per investigator)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.N. Roy Chengappa, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (4):
- United States (4):
  - Mayview State Hospital, Bridgeville, Pennsylvania
  - Dubois Regional Medical Center, DuBois, Pennsylvania
  - Mon-Yough Community Services, Inc., McKeesport, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Chengappa KN, Turkin SR, Schlicht PJ, Murphy SL, Brar JS, Fagiolini A, Houck PR, Garbutt RG, Fredrick N. A Pilot, 15-month, randomised effectiveness trial of Risperidone long-acting injection (RLAI) versus oral atypical antipsychotic agents (AAP) in persons with bipolar disorder. Acta Neuropsychiatr. 2010 Apr;22(2):68-80. doi: 10.1111/j.1601-5215.2010.00458.x. PMID 25385032

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone LAI: Oral Risperidone followed by Long acting Risperidone injections (Consta)
  Injectable Risperidone (Consta) or oral antipsychotic: Injectable Risperidone (Consta) from 12.5 to 50 mg q 2 weeks
- Oral AAP: Oral second generation antipsychotic agents other than clozapine or risperidone (olanzapine, quetiapine, ziprasidone, aripiprazole)
  Oral antipsychotic agents, olanzapine, quetiapine, ziprasidone, aripiprazole in doses approved in the US for bipolar disorder
Period: Overall Study
Arm/Group | Risperidone LAI | Oral AAP
Started | 23 | 25
Completed | 14 | 9
Not Completed | 9 | 16
Not completed — Protocol Violation | 0 | 7
Not completed — Lost to Follow-up | 4 | 5
Not completed — increase in alcohol and drug use | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — discharge from hospital | 1 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two patients in the Risperidone LAI group were not included in the analysis as they did not receive any assessment after the baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone LAI | Oral AAP | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — 2 patients in the risperidone LAI group were not included in the ITT (intention to treat) analyses as they did not receive assessment after the baseline assessment. Therefore, outcomes were assessed for only 23 of 25 patients in the risperidone LAI group.
  Participants
    Female | 16 | 18 | 34
    Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — 2 patients in the risperidone LAI group were not included in the ITT (intention to treat) analyses as they did not receive assessment after the baseline assessment. Therefore, outcomes were assessed for only 23 of 25 patients in the risperidone LAI group.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 3 | 9
    White | 16 | 22 | 38
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Number of Clinical Events (Pooled) Occurring Between 3-15 Months Following a Switch/Stabilization of the Antipsychotic Agents Among Patients Who Receive Either Risperidal Consta or One of the 4 Marketed 2nd Generation Antipsychotic Agents.
Time Frame: Upto 15 months
Population: 2 patients in the risperidone LAI group were not included in the ITT (intention to treat) analyses as they did not receive assessment after the baseline assessment. Therefore, outcomes were assessed for only 23 of 25 patients in the risperidone LAI group.
Measure: Mean (Standard Deviation); unit: Number of clinical events
Arm/Group | Risperidone LAI | Oral AAP
Number analyzed (Participants) | 23 | 25
Number of clinical events | 0.86 (0.73) | 1.61 (1.29)

2. Secondary Outcome: BMI
Description: BMI at baseline and at end of 15 months for Risperidone LAI and oral AAP groups
Time Frame: baseline to end of 15 months
Population: Patients with bipolar disorder
Measure: Mean (Standard Deviation); unit: kg / m^2
Arm/Group | Risperidone LAI | Oral AAP
Number analyzed (Participants) | 23 | 25
kg / m^2
  Baseline | 31.05 (7.20) | 29.86 (6.86)
  Final | 32.27 (8.31) | 32.0 (7.4)

3. Secondary Outcome: Number of Participants With Treatment - Emergent Hyperglycemia
Description: Number of participants with hyperglycemia based on safety labs
Time Frame: from baseline to end of 15 months
Population: patients with bipolar disorder
Measure: Number; unit: participants
Arm/Group | Risperidone LAI | Oral AAP
Number analyzed (Participants) | 23 | 25
participants | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Hyperlipidemia
Description: Number of participants with Hyperlipidemia as determined by safety labs
Time Frame: from baseline to end of 15 months
Population: patients with bipolar disorder
Measure: Number; unit: participants
Arm/Group | Risperidone LAI | Oral AAP
Number analyzed (Participants) | 23 | 25
participants | 0 | 0

ADVERSE EVENTS:
Description: 2 patients in the risperidone LAI group were not included in the ITT (intention to treat) analyses as they did not receive assessment after the baseline assessment. Therefore, outcomes were assessed for only 23 of 25 patients in the risperidone LAI group.
Arm/Group | Risperidone LAI | Oral AAP
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 23/23 | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone LAI (N=23) | Oral AAP (N=25)
Increased appetite (Metabolism and nutrition disorders) | 5 | 7
Somnolence (Nervous system disorders) | 6 | 4
Weight Gain (Metabolism and nutrition disorders) | 3 | 5
Migraine Headache (Nervous system disorders) | 4 | 3
tremors (Musculoskeletal and connective tissue disorders) | 4 | 2
Halucinations (Psychiatric disorders) | 0 | 4
Pain (Nervous system disorders) | 2 | 3
akathesia (Nervous system disorders) | 3 | 2
skin rash (General disorders) | 3 | 0
asthenia (General disorders) | 2 | 3
forgetfulness (Psychiatric disorders) | 2 | 2
URI (Respiratory, thoracic and mediastinal disorders) | 2 | 2
ademia (General disorders) | 2 | 1
dizziness (Nervous system disorders) | 1 | 2
constipation (Gastrointestinal disorders) | 2 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Menstrual distubances (Reproductive system and breast disorders) | 2 | 0
Lactation (Endocrine disorders) | 2 | 0
blurred vision (Eye disorders) | 0 | 2
heartburn (Gastrointestinal disorders) | 0 | 2
hyper glycemia (Endocrine disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No